CLINICAL TRIAL: NCT04907175
Title: Individual Patient Expanded Access IND to Evaluate the Safety and Efficacy of HB-adMSCs for the Treatment of Systemic Lupus Erythematosus (SLE)
Brief Title: Individual Patient Expanded Access IND of Autologous HB-adMSCs for the Treatment of Systemic Lupus Erythematosus (SLE)
Status: No longer available | Type: Expanded Access
Sponsor: Hope Biosciences Research Foundation (Industry)
Responsible Party: Sponsor
Other Study IDs: HBSLE01
Record Dates: First submitted 2021-05-26; First posted 2021-05-28 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: System; Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Biological: HB-adMSCs — Subject has completed 10 infusions and has been authorized for an additional 12 infusions over 1 year.
  Other Names: MSC's

SUMMARY:
This protocol is part of an FDA Individual Patient Expanded Access IND. This study is to be conducted according to US and International Standards of Good Clinical Practice (FDA Title 21 part 312 and International Conference on Harmonization guidelines), applicable government regulations and Hope Biosciences Stem Cell Research Foundation policies and procedures.

DETAILED DESCRIPTION:
This Individual Patient Expanded Access IND has been created per the request of a 65-year-old woman diagnosed with Systemic Lupus Erythematosus (SLE).

ELIGIBILITY:
Inclusion Criteria:

* Adult individual 18 years of age or older.
* Cognitively intact and capable of giving informed consent.
* Clinical diagnosis of Systemic Lupus Erythematosus.
* Subject has mesenchymal stem cells banked at Hope Biosciences.
* The patient accepts to receive treatment and to comply with follow-up visits.

Exclusion Criteria:

* Clinically significant, uncontrolled cardiovascular, lung, renal, hepatic, or endocrine diseases that in the opinion of the investigator may increase the risks associated with study participation.
* Active Alcohol or Drug addiction.
* Participation in concurrent interventional research studies during this study.
* Severe organ failure (heart, kidney or liver) confirmed by additional tests or medical history.
* Unwillingness to return for follow-up visits.

Ages: 18 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Thanh Cheng, MD, Principal Investigator — Hope Biosciences Stem Cell Research Foundation
Locations (1):
- Hope Biosciences Stem Cell Research Foundation, Sugar Land, Texas, United States